CLINICAL TRIAL: NCT04612101
Title: Checking Brain Temperature Through MRI Thermometry
Brief Title: Check Brain Temp Trial
Status: Completed | Type: Observational
Sponsor: OSF Healthcare System (Other)
Collaborators: University of Illinois College of Medicine at Peoria (Other)
Responsible Party: Principal Investigator, WenChing Liu, Clinical Medical Physicist, OSF Healthcare System
Other Study IDs: 1140816
Record Dates: First submitted 2020-10-27; First posted 2020-11-02 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: the Focus of the Clinical Trial is on the Brain Temperatures in Normal Human Subjects
Keywords: MR Thermometry; Human brain temperature; MR spectroscopy; normal brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite some controversial results, many patients and animal studies have suggested significant benefit of using hypothermia treatment in stroke patient population. However, certain questions for how to applying this therapy properly such as when to start, what is the optimal temperature, how long is the duration, and what is the best hypothermia technology that may avoid the complications including focal soft tissue injuries are still remain questioned.

In this study, we will utilize the linear relationship of temperature vs. chemical shift in MR Spectroscopy to measure the brain temperatures in normal men.

DETAILED DESCRIPTION:
Brain temperature has an interactive relationship with brain cell metabolism. Hypothermia is a known neuronal protectant therapy. It has been proven to be effective in reducing the brain injury in patients post cardiac arrest. However, the role of hypothermia in brain or spinal cord injury such as in either hemorrhagic or ischemic condition remains unclear. Many questions on hypothermia are unanswered. For example, what is the optimal low temperature in order to have the maximum therapeutic effect? How long should hypothermia be applied for? Is there a regional temperature difference between different parts of brain in physiological or pathological conditions? In order to answer these questions, the first step is to have a reliable way of measuring brain temperature accurately. However, invasive technique such as inserting temperature probe to different parts of brain is not practical. Using body core temperature to estimate the intracranial temperature is inaccurate.

To establish a noninvasive means to obtain and monitor brain temperature in a dynamic environment is the essential step in order to studying hypothermia and answering the questions mentioned earlier. MRI brain thermometry is a fast, direct and non-invasive method to estimate the brain temperature with great accuracy. This technique is based on several temperature dependent physical properties in our brain such as chemical shift between metabolites and water. Currently, there is no standard MRI brain thermometry in physiological and pathological conditions such as stroke. We plan to explore and establish MRI brain thermometry. The first step is to establish temperature correlation on measured water temperature.

Then temperature of different regions of brain will be used to compare to the standardized water temperature in normal people.

ELIGIBILITY:
Inclusion Criteria:

* Normal and healthy

Exclusion Criteria:

* 1. claustrophobia, 2. history of neurological disease. 3. Tattoo and 4. History of lost conscience due to any head injury.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: normal and healthy Men
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Brian temperatures | Brain temperatures were taken during an hour
  Brian temperatures were measured at region of interests

CONTACTS AND LOCATIONS:
Locations (1):
- OSF Healthcare Saint Francis Medical Center, Peoria, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided